CLINICAL TRIAL: NCT04231344
Title: Prevalence of Laryngeal Disorders in Patients With GERD in Assiut University Hospital
Brief Title: Laryngeal Disorders and GERD in Assiut University
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SHimaa Salah Sadek, Principle investigator, Assiut University
Other Study IDs: LPRD
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Laryngeal Disease
MeSH Terms: conditions — Laryngeal Diseases | interventions — Laryngoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Laryngoscopy — Laryngoscopic examination of patients with GERD by two physicians

SUMMARY:
Study laryngeal disorders by laryngoscopic examination by two physicians on GERD patients diagnosed by gastroenterology department by endoscopy and effect of GERD treatment for 3 months on these laryngeal disorders without any treatment to laryngeal disorders

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed GERD by gastroenterology department before start of treatment and have laryngeal symptoms

Exclusion Criteria:

* voice abusers as singers ,teachers and readers.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who diagnosed GERD by gastroenterology department before start of treatment of GERD Will examine by laryngoscopy for laryngeal lesions then they Will take treatment to GERD by gastroenterology department without any treatment to laryngeal disorders and study effect of GERD treatment on these laryngeal disorders
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of laryngeal disorders in GERD patients | One year from February 2020 to February 2021
  Laryngoscopic examination of patients with GERD by two otorhinolaryngologist physicians

SECONDARY OUTCOMES:
Effect of treatment of GERD on these laryngeal disorders | 3 months
  Treatment of GERD by gastroenterology department for 3 months and reexamination of patients by laryngoscopy for laryngeal disorders without any treatment to laryngeal disorders

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Cohen JT, Bach KK, Postma GN, Koufman JA. Clinical manifestations of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):19-23. PMID 12353427
- [Background] Belafsky PC, Postma GN, Amin MR, Koufman JA. Symptoms and findings of laryngopharyngeal reflux. Ear Nose Throat J. 2002 Sep;81(9 Suppl 2):10-3. PMID 12353425